CLINICAL TRIAL: NCT00799162
Title: Prediction of Post-Cesarean Section Pain
Acronym: PPCSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ruth Landau, Professor, University of Washington
Other Study IDs: 35115-A
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women with a scheduled cesarean section
  Interventions: Other: Psychophysical testing, questionnaires, and genetics

INTERVENTIONS:
Other: Psychophysical testing, questionnaires, and genetics — pre-operative psychophysical testing of endogenous pain modulation, pre-operative questionnaires, peri- and post-operative data collection, long term follow-up assessing chronic pain, SNP association analysis, and whole genome scanning association studies

SUMMARY:
The purpose of this study is to determine if dynamic psychophysical testing along with genetic screening will allow to identify pre-operatively women who will suffer severe acute pain post-operatively and the subset who may experience chronic pain following cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-50 scheduled for an elective cesarean section (1st or 2nd cesarean section)

Exclusion Criteria:

Women who:

* have taken opioids, acetaminophen, or NSAIDs 48 hrs prior to psychophysical testing
* have had more than two previous cesarean sections
* have a vertical abdominal incision from a prior cesarean section
* are non-English speaking
* have mental health issues
* have a failure of spinal anesthetic and require conversion to general anesthesia
* have a vertical uterine incision performed during ongoing cesarean section
* have a previous vertical uterine scar discovered during ongoing cesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with a scheduled elective cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Stanford University, Stanford, California
  - University of Washington, Seattle, Washington
- St. Luc Hospital, University Catholic of Louvain, Brussels, Brussels Capital, Belgium
- Hospital e Maternidade Santa Joana, São Paulo, São Paulo, Brazil
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Ortner CM, Turk DC, Theodore BR, Siaulys MM, Bollag LA, Landau R. The Short-Form McGill Pain Questionnaire-Revised to evaluate persistent pain and surgery-related symptoms in healthy women undergoing a planned cesarean delivery. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):478-86. doi: 10.1097/AAP.0000000000000158. PMID 25304476